CLINICAL TRIAL: NCT07017985
Title: Prevalence of Diabetes in Patients Who Are Candidates for Spine Surgery
Acronym: PREDIR
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-06-007
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Spine Disease
Keywords: Spine surgery; Diabetes
MeSH Terms: conditions — Spinal Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to assess, through systematic screening, the prevalence of diabetes or prediabetes in patients who are candidates for lumbar spine surgery.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, single-center, open-label observational study on a population of patients undergoing lumbar spine surgery.

This study does not alter patient management or the physician-patient relationship. Assessments take place during routinely scheduled consultations. Fasting blood glucose and glycated hemoglobin measurements are part of the standard preoperative assessment. Patient self-administered questionnaires are routinely completed for practice evaluation purposes and constitute a database for routine care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients,
* Patients who have been informed of the research and have not indicated their opposition to the use of their medical data,
* Patients who are candidates for their first lumbar spine surgery, whether instrumented or not

Exclusion Criteria:

* Non-instrumented percutaneous surgery (cementoplasty)
* Presence of spinal osteosynthesis equipment
* Surgery performed for an infectious or tumoral spinal condition
* Surgery via an anterior or lateral approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of patients who are candidates for lumbar spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Diabetes or prediabetes présence | Day 1
  Diabetes is defined as a blood glucose level of at least 1.26 g/L and a glycated hemoglobin level greater than or equal to 6.5%.
  Prediabetes is defined as a blood glucose level greater than 1.10 g/L and less than 1.26 g/L and a glycated hemoglobin level between 5.7% and 6.4%.

SECONDARY OUTCOMES:
Low back pain | Day 0
  Pain will be assessed by the patient on a visual analog scale from 0 to 10 (0 = no pain, 10 = maximum pain).
Low back pain | Month 3
  Pain will be assessed by the patient on a visual analog scale from 0 to 10 (0 = no pain, 10 = maximum pain).
Radicular pain | Day 0
  Pain will be assessed by the patient on a visual analog scale from 0 to 10 (0 = no pain, 10 = maximum pain).
Radicular pain | Month 3
  Pain will be assessed by the patient on a visual analog scale from 0 to 10 (0 = no pain, 10 = maximum pain).
Functional Impact of the Disease | Day 0
  Functional Impact of the Disease is assessed with the Oswestry Disability Index (ODI) questionnaire. The ODI questionnaire consists of 10 questions regarding: pain, self-care, lifting, walking, sitting, standing, sleeping, sexual activity, social activity, and traveling. Each question offers six answers, with a score from 0 to 6, for the patient to select; a score of 0 corresponds to normal function, and a score of 6 to very impaired function. The resulting score is multiplied by 2 to obtain a percentage of disability, with 0% indicating no disability and 100% indicating the most significant disability. A score between 0 and 20% indicates minimal disability, a score between 21 and 40% indicates moderate disability, a score between 41 and 60% indicates severe disability, and a score above 61% indicates major disability.
Functional Impact of the Disease | Month 3
  Functional Impact of the Disease is assessed with the Oswestry Disability Index (ODI) questionnaire. The ODI questionnaire consists of 10 questions regarding: pain, self-care, lifting, walking, sitting, standing, sleeping, sexual activity, social activity, and traveling. Each question offers six answers, with a score from 0 to 6, for the patient to select; a score of 0 corresponds to normal function, and a score of 6 to very impaired function. The resulting score is multiplied by 2 to obtain a percentage of disability, with 0% indicating no disability and 100% indicating the most significant disability. A score between 0 and 20% indicates minimal disability, a score between 21 and 40% indicates moderate disability, a score between 41 and 60% indicates severe disability, and a score above 61% indicates major disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jacques Cartier, Massy, France